CLINICAL TRIAL: NCT01664767
Title: Placebo Controlled Study Evaluating the Modulatory Effects of Sulfur Thermal Water Inhalation on Superoxide Anion Levels in Exhaled Breath Condensate in COPD Patients
Brief Title: Effects of Sulfur Thermal Water Inhalation on Airway Oxidative Stress in COPD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi di Ferrara (Other)
Collaborators: Terme di Riolo Spa (Unknown)
Responsible Party: Principal Investigator, Alberto Papi, MD, Professor, Università degli Studi di Ferrara
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTUNIFE01
Record Dates: First submitted 2012-08-10; First posted 2012-08-14 (Estimated); Last update posted 2013-12-30 (Estimated); Status verified 2013-12

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; Thermal water; Oxidative stress; Inflammation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Thermal water inhalation (Experimental): Patients will perform 12 days of sulfur thermal water inhalation
  Interventions: Other: Sulfur Thermal water
- Isotonic saline inhalation (Placebo Comparator): Patients will perform 12 days of isotonic saline inhalation
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Sulfur Thermal water
  Arms: Thermal water inhalation
Other: Placebo
  Arms: Isotonic saline inhalation

SUMMARY:
The chronic obstructive pulmonary disease (COPD) is a chronic inflammatory disease of the airways characterized by fixed airflow obstruction, with important systemic co-morbidities. The obstruction is usually progressive and irreversible despite chronic therapy. Cigarette smoking is the major cause of this disease. COPD is an important cause of morbidity and mortality worldwide. Numerous studies have shown that oxidative stress plays a key role in the pathogenesis of COPD. In particular, the active metabolites of oxygen such as superoxide anion and the hydroxyl radical are unstable molecules that can trigger significant oxidative processes at the cellular level. These molecules can alter the extracellular matrix remodeling, cell respiration, cell proliferation, cellular repair and the immune response in the lung. All these events are key elements in the pathogenesis of COPD.

Currently available treatments for COPD (i.e. long-acting bronchodilators and inhaled corticosteroids) have not demonstrated a significant in vivo antioxidant effect. The thermal inhalation treatments are a therapeutic strategy used since many years in an empirical way in patients with COPD. Indeed, the evidence of effectiveness of spa treatment in patients with COPD are very limited.

The aim of this in vivo study is to evaluate the modulatory effects of sulfur thermal water inhalation on oxidant stress in the airways of stable COPD patients.

ELIGIBILITY:
Inclusion Criteria:

* Forty stable moderate to severe COPD patients (Global Initiative for Chronic Obstructive Lung Disease (GOLD) stage 2 and 3), according to international guidelines.
* FEV1/FVC ratio post-bronchodilator <70%
* 30% < FEV1 < 80%

Exclusion Criteria:

* Atopy
* Asthma
* Concomitant lung diseases (e.g. lung cancer)
* Acute infections of the respiratory tree in the previous 3 months including COPD exacerbation.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-11; Primary Completion 2013-01 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Superoxide anion levels in exhaled breath condensate | 12 days
  Levels of superoxide anion levels will be measured at recruitment (day 0) and after 12 days of inhalation. Changes between day 12 and day 0 will be evaluated.

SECONDARY OUTCOMES:
Superoxide anion levels in exhaled breath condensate | 42 day
  Levels of superoxide anion will be measured at recruitment (day 0), after 12 days of inhalation (day 12) and one month after the last day oh inhalation (day 42). Changes between day 42, day 12 and day 0 will be evaluated.
Inflammatory cell counts in induced sputum | 42 days
  Inflammatory cell counts in induced sputum will be measured at recruitment (day 0), after 12 days of inhalation (day 12) and one month after the last day of inhalation (day 42). Changes between day 42, day 12 and day 0 will be evaluated.
Clinical outcomes | 42 days
  Spirometry and the impact of COPD on patient quality of life (performed by the COPD Assessment Test (CAT)) will be measured at recruitment (day 0), after 12 days of inhalation (day 12) and one month after the last day of inhalation (day 42). Changes between day 42, day 12 and day 0 will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Centre on Asthma and COPD, University of Ferrara, Ferrara, Italy

REFERENCES:
- [Derived] Contoli M, Gnesini G, Forini G, Marku B, Pauletti A, Padovani A, Casolari P, Taurino L, Ferraro A, Chicca M, Ciaccia A, Papi A, Pinamonti S. Reducing agents decrease the oxidative burst and improve clinical outcomes in COPD patients: a randomised controlled trial on the effects of sulphurous thermal water inhalation. ScientificWorldJournal. 2013 Dec 23;2013:927835. doi: 10.1155/2013/927835. eCollection 2013. PMID 24453924